CLINICAL TRIAL: NCT03503617
Title: RehabTouch: A Mixed-reality Gym for Rehabilitating the Hands, Arms, Trunk, and Legs After Stroke
Brief Title: RehabTouch Home Therapy for Stroke Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Flint Rehabilitation Devices, LLC (Industry)
Collaborators: Rancho Research Institute, Inc. (Other)
Responsible Party: Principal Investigator, Flint Rehabilitation Devices, LLC, Vice President, Flint Rehabilitation Devices, LLC
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 1R44AG059256-01A1 (NIH)
Record Dates: First submitted 2018-04-11; First posted 2018-04-20 (Actual); Results first posted 2022-02-07 (Actual); Last update posted 2022-02-07 (Actual); Status verified 2022-01

CONDITIONS: Cerebral Stroke
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (2):
- RehabTouch Exercise Program (Experimental): Participants will perform targetted movement exercises by interacting with the RehabTouch pucks, as described and monitored on a computer. Participants will be asked to exercise at least 3 hours per week for 3 consecutive weeks.
  Interventions: Device: RehabTouch
- Conventional tabletop exercise program (Active Comparator): Conventional tabletop exercise program is a traditional exercise program described in a booklet similar to what is typical provided to stroke patients upon their discharge from the hospital. Participants will be asked to perform these exercises at least 3 hours per week for 3 consecutive weeks.
  Interventions: Other: Conventional tabletop exercise program

INTERVENTIONS:
Device: RehabTouch — Exercise using the motion sensing devices and a computer
  Other Names: FitMi
  Arms: RehabTouch Exercise Program
Other: Conventional tabletop exercise program — Exercise following printed sheets of exercises
  Arms: Conventional tabletop exercise program

SUMMARY:
We will investigate the efficacy of a newly developed exercise device (RehabTouch) for people in the subacute stage after a stroke compared to a traditional tabletop exercise program. RehabTouch uses embedded sensors that can track and record the patient's direction and degree of movement as they perform exercises described on a computer.

ELIGIBILITY:
Inclusion Criteria:

* Age: 18 to 85 years old
* Upper extremity weakness measured by a clinical scale
* Absence of moderate to severe pain on affected upper extremity
* Able to understand the instructions to operate RehabTouch

Exclusion Criteria:

* Concurrent severe medical problems, visual deficits, severe neglect or apraxia
* Enrollment to other therapy studies

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 27 (Actual)
Dates: Start 2018-11-01 (Actual); Primary Completion 2021-03-31 (Actual); Study Completion 2021-03-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Susan Shaw, MD, Principal Investigator — Rancho Research Institute, Inc.
Locations (1):
- Rancho Research Institute, Inc., Downey, California, United States

REFERENCES:
- [Derived] Swanson VA, Johnson C, Zondervan DK, Bayus N, McCoy P, Ng YFJ, Schindele Bs J, Reinkensmeyer DJ, Shaw S. Optimized Home Rehabilitation Technology Reduces Upper Extremity Impairment Compared to a Conventional Home Exercise Program: A Randomized, Controlled, Single-Blind Trial in Subacute Stroke. Neurorehabil Neural Repair. 2023 Jan;37(1):53-65. doi: 10.1177/15459683221146995. Epub 2023 Jan 12. PMID 36636751

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | RehabTouch Exercise Program | Conventional Tabletop Exercise Program
Started | 14 | 13
Completed | 14 | 10
Not Completed | 0 | 3

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | RehabTouch Exercise Program | Conventional Tabletop Exercise Program | Total
Number analyzed (Participants) | 14 | 13 | 27
Age, Continuous [Mean (Standard Deviation); unit: Years] | 50 (11) | 52 (9) | 52 (10)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 4 | 4
  Male | 14 | 9 | 23
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 8 | 10 | 18
  Not Hispanic or Latino | 6 | 3 | 9
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 2 | 1 | 3
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 2 | 3
  White | 1 | 2 | 3
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 10 | 8 | 18
Region of Enrollment [Number; unit: participants]
  United States | 14 | 13 | 27

OUTCOME MEASURES:

1. Primary Outcome: Change in Fugl-Meyer Arm Motor Score From Baseline to One Month Post Therapy
Description: The Fugl-Meyer Arm Motor Score is a stroke-specific, performance-based impairment index which measure 33 arm movement patterns based on a scale of 0 to 2 each, for a total possible score of 66. For each movement patter, a score of zero means the participant is unable to perform the movement pattern; a score of 2 means the participant performed the movement patterns faultlessly.
Time Frame: From Baseline to One-month Post-therapy
Population: Three participants in the conventional therapy group did not perform their one-month follow-up assessment; one of these did perform the end-of-therapy assessment. For this one participant, the missing one-month follow-up data point was imputed for the primary outcome measure by adding the average change in Fugl-Meyer score across all participants in the conventional therapy group from end-of-therapy to one-month follow-up to this participant's end-of-therapy Fugl-Meyer score.
Measure: Mean (Standard Deviation); unit: Score on a Scale
Arm/Group | RehabTouch Exercise Program | Conventional Tabletop Exercise Program
Number analyzed (Participants) | 14 | 11
Score on a Scale | 8.0 (4.6) | 3.1 (6.1)
Statistical Analysis 1: Comparison: RehabTouch Exercise Program vs Conventional Tabletop Exercise Program; Test type: Superiority; p = 0.03, t-test, 2 sided

2. Secondary Outcome: Change in Box and Blocks Test Score
Description: The Box & Blocks Test (BBT) score assess hand function and gripping ability by instructing an individual to move as many blocks as possible, one at a time, from one compartment to the other for a period of 60 seconds. The BBT is scored by counting the number of blocks carried over the partition from one compartment to the other during the one-minute trial period.
Time Frame: From Baseline to One-month Post-therapy
Measure: Mean (Standard Deviation); unit: Boxes
Arm/Group | RehabTouch Exercise Program | Conventional Tabletop Exercise Program
Number analyzed (Participants) | 14 | 10
Boxes | 31.1 (20.2) | 27.1 (16.9)

3. Secondary Outcome: 10 Meter Walk Test
Description: The 10MWT assesses walking speed in meters per second over a short duration.
Time Frame: From Baseline to One-month Post-therapy
Measure: Mean (Standard Deviation); unit: meters per second
Arm/Group | RehabTouch Exercise Program | Conventional Tabletop Exercise Program
Number analyzed (Participants) | 14 | 10
meters per second | 1.06 (0.41) | 1.07 (0.39)

4. Secondary Outcome: Motor Activity Log
Description: The Motor Activity Log (MAL) is a semi-structured interview to assess arm function after hemiparetic stroke. Individuals are asked to rate Quality of Movement (QOM) and Amount of Movement (AOM) during 28 daily functional tasks on a 0-5 point scale. For the QOM subscale, 0 represents an inability to use the affected arm to perform an activity, while 5 represents a normal ability to use the affected arm. For the AOM scale, 0 represents never using the affected arm to perform the activity, and 5 indicates always using the affected arm to perform the activity.
Time Frame: One-month Post-therapy
Measure: Mean (Standard Deviation); unit: Score on a Scale
Arm/Group | RehabTouch Exercise Program | Conventional Tabletop Exercise Program
Number analyzed (Participants) | 14 | 10
Score on a Scale
  Amount of Use | 3.11 (1.14) | 2.72 (1.65)
  How Well | 3.01 (1.26) | 2.50 (1.53)

5. Secondary Outcome: Visual Analog Pain Scale
Description: A standard analog scale that ranges from 0 to 10 for assessing pain.
Time Frame: From Baseline to One-month Post-therapy
Measure: Mean (Standard Deviation); unit: Score on a Scale
Arm/Group | RehabTouch Exercise Program | Conventional Tabletop Exercise Program
Number analyzed (Participants) | 14 | 10
Score on a Scale | 2.5 (2.3) | 4.6 (3.1)

6. Secondary Outcome: Modified Ashworth Spasticity Scale
Description: The Modified Ashworth Spasticity (MAS) Scale measures spasticity in patients with lesions of the Central Nervous System. Tests resistance to passive movement about a joint with varying degrees of velocity, with movements in flexion and extension scored separately. Scores for each movement direction and joint range from 0-5, with 6 choices. A score of 0 indicates no increase in tone during movement. A score of 5 indicates that the limb was rigid during the passive movement.
Time Frame: From Baseline to One-month Post-therapy
Measure: Mean (Standard Deviation); unit: Score on a Scale
Arm/Group | RehabTouch Exercise Program | Conventional Tabletop Exercise Program
Number analyzed (Participants) | 14 | 10
Score on a Scale
  Extension | 0.42 (0.7) | 0.63 (0.92)
  Flexion | 2.5 (2.1) | 2.1 (2.3)

ADVERSE EVENTS:
Time Frame: 1 year, 4 months
Arm/Group | RehabTouch Exercise Program | Conventional Tabletop Exercise Program
All-Cause Mortality (participants affected / at risk) | 0/14 | 0/13
Serious Adverse Events (participants affected / at risk) | 0/14 | 0/13
Other Adverse Events (participants affected / at risk) | 0/14 | 0/13

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-08-31): https://cdn.clinicaltrials.gov/large-docs/17/NCT03503617/Prot_SAP_002.pdf